CLINICAL TRIAL: NCT00260754
Title: Utilization of the Community Popular Opinion Leader (C-POL) Model to Achieve Syphilis Elimination in Alabama
Brief Title: Utilization of the Community Popular Opinion Leader (C-POL) Model in Alabama
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4087; U65/CCU422269
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2006-05-31 (Estimated); Status verified 2005-12

CONDITIONS: Risk Behavior; Sexually Transmitted Diseases
Keywords: Risk behavior; Sexually transmitted diseases
MeSH Terms: conditions — Risk-Taking; Sexually Transmitted Diseases

INTERVENTIONS:
Behavioral: Community-Popular Opinion Leader Model
Behavioral: Diffusion of Innovations

SUMMARY:
Community members within the treatment city will report: 1)engaging in fewer sexual risk practices; 2)significantly higher condom use; 3) significantly higher rates of STD care seeking (including STD screening behaviors); 4) fewer having STDs in the past 6 months; 5) significantly higher awareness scores regarding syphilis and other STDs, as compared with those in the comparison city.

DETAILED DESCRIPTION:
The C-POL in Alabama project is and intervention study which sought to impact the health behaviors of community residents who live in zip codes that have high syphilis morbidity. The study is being implemented in Birmingham and Montgomery with shelter clients.

The intervention model used for this study is the Popular Opinion Leader (POL) model, which is effective at reducing new HIV infections. The intent of this study was to determine the effectiveness of a diffusion model (e.g. POL) at reducing syphilis infections in affected communities.

For the intervention, community members identified as popular opinion leaders were recruited and trained to share accurate information about syphilis transmission, symptoms, testing, treatment and prevention. Prior to intervention implementation and several times after, community members were given a survey and screened for syphilis as well as 2-3 additional STDs. During each assessment, cross-sections of the community members were sampled.

ELIGIBILITY:
Inclusion Criteria:

* Clients who utilized two community homeless shelters in the affected community. The affected community was one that had significant syphilis morbidity at the onset of the study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-10; Study Completion 2005-07

PRIMARY OUTCOMES:
Changes in syphilis morbidity in affected community

SECONDARY OUTCOMES:
Changes in risk behavior and health care seeking behavior

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Williams, Ph.D., Study Chair — CDC/NCHSTP/DSTDP/BIRB; Diane Grimley, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Birmingham, Alabama, United States